CLINICAL TRIAL: NCT04213430
Title: Development and Validation of a Deep Learning System for Multiple Ocular Fundus Diseases Using Retinal Images: a Multi-center Prospective Study
Brief Title: Development and Validation of a Deep Learning System for Multiple Ocular Fundus Diseases Using Retinal Images
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Prof., Sun Yat-sen University
Other Study IDs: CCPMOH2019- China8
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Ophthalmological Disorder
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training dataset: Retinal images collected from hospitals and multiple screening sites all over China
- Validation dataset: Retinal images separated from training dataset
  Interventions: Other: diagnostic
- Testing dataset: Retinal images prospectively collected from the hospitals and ocular disease screening sites totally different from training dataset
  Interventions: Other: diagnostic

INTERVENTIONS:
Other: diagnostic — Training dataset was used to train the deep learning model, which was validated and tested by other two datasets.
  Groups: Testing dataset; Validation dataset

SUMMARY:
Retinal images can reflect both fundus and systemic conditions (diabetes and cardiovascular disease) and firstly to be used for medical artificial intelligence (AI) algorithm training due to its advantages of clinical significance and easy to obtain. Here, the investigators developed a single network model that can mine the characteristics among multiple fundus diseases, which was trained by plenty of fundus images with one or several disease labels (if they have) in each of them. The model performance was compared with those of both native and international ophthalmologists. The model was further tested by datasets with different camera types and validated by three external datasets prospectively collected from the clinical sites where the model would be applied.

ELIGIBILITY:
Inclusion Criteria:

* The quality of fundus images should clinical acceptable. More than 80% of the fundus image area including four main regions (optic disk, macular, upper and lower retinal vessel archs) are easy to read and discriminate.

Exclusion Criteria:

* Images with light leakage (>30% of area), spots from lens flares or stains, and overexposure were excluded from further analysis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Retinal images were collected from different health care institutes all over China and other countries around the world.
Sampling Method: Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve of the deep learning system | baseline
  The investigators will calculate the area under the receiver operating characteristic curve of deep learning system and compare this index between deep learning system and human doctors.

SECONDARY OUTCOMES:
Sensitivity of the deep learning system | baseline
  The investigators will calculate the sensitivity of deep learning system and compare this index between deep learning system and human doctors.
Specificity of the deep learning system | baseline
  The investigators will calculate the specificity of deep learning system and compare this index between deep learning system and human doctors.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin D, Xiong J, Liu C, Zhao L, Li Z, Yu S, Wu X, Ge Z, Hu X, Wang B, Fu M, Zhao X, Wang X, Zhu Y, Chen C, Li T, Li Y, Wei W, Zhao M, Li J, Xu F, Ding L, Tan G, Xiang Y, Hu Y, Zhang P, Han Y, Li JO, Wei L, Zhu P, Liu Y, Chen W, Ting DSW, Wong TY, Chen Y, Lin H. Application of Comprehensive Artificial intelligence Retinal Expert (CARE) system: a national real-world evidence study. Lancet Digit Health. 2021 Aug;3(8):e486-e495. doi: 10.1016/S2589-7500(21)00086-8. PMID 34325853